CLINICAL TRIAL: NCT00648986
Title: Single Center, Open-Label, Efficacy and Safety Study of Tazarotene (Tazorac) for the Treatment of Brittle Nails
Brief Title: Efficacy and Safety Study of Tazarotene (Tazorac) for the Treatment of Brittle Nails
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Richard K. Scher, M.D./Principal Investigator, Columbia University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA5735; TAZ11-2003 (Other: Allergan)
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Brittle Nails
Keywords: brittle nails; Tazarotene; Tazorac
MeSH Terms: conditions — Twenty-Nail Dystrophy | interventions — tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Uncontrolled, Open-Label Pilot Study
  Interventions: Drug: Tazorac

INTERVENTIONS:
Drug: Tazorac — All patients were to apply topical tazarotene (Tazorac) twice daily to all affected fingernails for 24 weeks.
  Other Names: Tazarotene

SUMMARY:
The purpose of this study is to determine whether topical tazarotene (Tazorac), a receptor-selective synthetic retinoid that normalizes epidermal differentiation, ameliorates signs and symptoms of brittle nails.

DETAILED DESCRIPTION:
"Brittle nails," referring to nails that chip, peel, or split excessively, occur in up to 30% of women and 15% of men, with highest prevalence among the elderly. Treatment of brittle nails involves restoration and maintenance of a normal degree of nail plate hydration by minimizing exposure to dehydrating chemicals and by use of moisturizers, such as alpha-hydroxy acids. Retinoids are vitamin A analogs that play a role in skin cell differentiation and proliferation. Tazarotene is a topical receptor-selective synthetic retinoid that normalizes epidermal differentiation and reduces the influx of inflammatory cells into the skin. In this single-center, open-label trial, subjects applied tazarotene to the nails twice daily for 24 weeks. Signs and symptoms were rated by the investigators and subjects during treatment and 12 weeks after discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided IRB-approved written informed consent prior to conducting any study-related procedures
* Men and female patients 18 to 75 years of age
* Have had a diagnosis of brittle nails
* Have two target fingernails identified at baseline
* Have evidence of at least two of the following signs and symptoms of brittle nails in each of the selected nail plates or severe signs (one or more) on each target nail:
* trachyonychia (surface roughness)
* lamellar onychoschizia (horizontal layering)
* longitudinal cracking or splitting of the distal edge
* Female patient of childbearing potential (not surgically sterile or at least 2 years postmenopausal) has a negative pregnancy test at baseline/day 1 and is not lactating
* Sexually active female subject who is not surgically sterile or 2 years post menopausal must agree to use contraception/birth control measure while on study (e.g., oral contraceptives, diaphragms with spermicide, condoms with spermicide, intrauterine devices, Norplant System, Depo-Provera, tubal ligation)
* Patients will agree to self-administer topical study medication, and will agree to complete all study procedures
* Patient is judged to be in good health by medical history and physical examination
* Must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Have a history of surgery of the affected fingernails
* Are pregnant, nursing, or planning pregnancy prior to study enrollment
* Have a disturbance of the shape of the affected fingernails (e.g., due to malformation of the underlying bone) that would interfere with the investigator's ability to evaluate photographs
* Have onycholysis (lifting of the nail plate off the nailbed) of the affected fingernails
* Have a fungal infection of the affected fingernails
* Have a history of psoriasis or lichen planus involving any nail, or active contact dermatitis involving the affected fingernails
* Have used any topical cosmetics or medicated products on the affected nails within 2 weeks of baseline visit
* Have received oral antifungal treatment within 3 months of baseline visit
* Have a known or suspected history of a genetic condition affecting the nails (e.g., Darier's disease, nail-patella syndrome, tuberculosis sclerosis)
* Immune compromise due to HIV infection, organ transplantation, or treatment of malignancy
* Chronic liver, heart, kidney, or ( untreated) thyroid disease
* Have used any investigational drug within the previous 1 month or 5 half-lives of the investigational agent, whichever is longer, or 3 months for any biologic of unknown half-life
* Are known to have had a substance abuse (drug or alcohol) problem within the previous 3 years
* Unlikely to comply with the study protocol and prescribed treatment or is unsuitable for any other reason in the opinion of the investigator
* Have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease;
* Currently have any known malignancy or have a history of malignancy other than non-melanoma skin cancer
* Are known to be infected with human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Have signs of bacterial, fungal or viral skin lesions that may interfere with measurement of the target lesions.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the change in the Physician's Global Improvement Assessment (PGIA) of the 2 target nails. The PGIA score reflects the comparison of photographs taken at baseline to the nails at 12 weeks, 24 weeks, and 36 weeks. | Weeks 12, 24, and 36

SECONDARY OUTCOMES:
Physician's Global Assessment (PGA) measures the severity of brittle nail symptoms. | Baseline, Week 12, and Week 24
Physician ratings of the roughness, raggedness, and peeling of the target nails. | All study visits
A VapoMeter measures the Transonychial Water Loss (TOWL) on both target nails. | All study visits
Subject reporting provides the subjects' assessments of their nail breakage. | All study visits
Subject reporting provides the subjects' satisfaction with the product. | Week 12, 24, and 36

CONTACTS AND LOCATIONS:
Overall Officials: Richard Scher, MD, Principal Investigator — University of North Carolina; Julian Mackay-Wiggan, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States